CLINICAL TRIAL: NCT06769880
Title: Combating Health Disparities Using Bedside Imaging and Community Health Workers for Early Screening and Referral of Pre-symptomatic Stage B Heart Failure in the Emergency Department
Brief Title: Use of Bedside Imaging and Community Health Workers for Early Screening and Referral of Pre-symptomatic Stage B Heart Failure in the Emergency Department
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Michael Gottlieb, Professor of Emergency Medicine, Vice Chair of Research, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23112905; P50MD017349 (NIH)
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Heart Diseases
Keywords: POCUS; Ultrasound; Ultrasonography; Echocardiography
MeSH Terms: conditions — Heart Diseases | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Intervention Alone (Placebo Comparator)
  Interventions: Other: Educational Intervention Alone
- Ultrasound and Educational Intervention (Experimental)
  Interventions: Other: Ultrasound and Educational Intervention

INTERVENTIONS:
Other: Ultrasound and Educational Intervention — This will include the educational intervention combined with a point-of-care ultrasound
  Arms: Ultrasound and Educational Intervention
Other: Educational Intervention Alone — This will include only the educational intervention (without ultrasound)
  Arms: Educational Intervention Alone

SUMMARY:
The goal of this clinical trial is to learn if using point-of-care ultrasound (POCUS) can increase participant engagement and changes in behavior among adults with risk factors for pre-symptomatic heart failure presenting to the emergency department. The main questions it aims to answer are:

1. Does POCUS increase understanding of heart failure and the likelihood to improve diet, exercise, and follow up?
2. Does POCUS improve diet, exercise, follow up, and self-efficacy at three months post-intervention?

Researchers will compare an educational intervention with versus without POCUS to see if POCUS works to improve outcomes.

Participants will:

Receive either the educational intervention alone or an educational intervention plus POCUS. They will report the difference in their understanding and likelihood to improve diet, exercise, and follow up immediately post-intervention. They will also report changes in diet, exercise, follow up, and self-efficacy at three months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Must be 45 years of age or older
* Must have high blood pressure, diabetes mellitus, or obesity (body mass index ≥30 kg/m2)

Exclusion Criteria:

* Symptoms of acute heart failure (difficulty breathing, leg swelling)
* History of heart failure
* Unable to tolerate an ultrasound examination
* No access to a phone for follow up

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Primary Care Follow Up | 3 Months Post-Intervention
  Defined as the presence or absence of a follow up visit with a primary care provider at 3 months

SECONDARY OUTCOMES:
Likelihood to Follow Up with a Primary Care Physician within the 3 Months Post-Intervention | Baseline and Immediately Post-Intervention
  Ordinal scale of 1 (very unlikely) to 7 (very likely)
Self-perceived knowledge of heart failure | Baseline and Immediately Post-Intervention
  Ordinal scale of 1 (no knowledge) to 7 (extremely knowledgeable)
Degree of motivation and self-efficacy using a modified High Blood Pressure Self-Care Profile (HBP-SCP) Motivation and Self-Efficacy tool | Baseline, Immediately Post-Intervention, and 3 Months Post-Intervention
Likelihood to change their fruit and vegetable intake using the Stages of Change tools for Fruits and Vegetables | Baseline, Immediately Post-Intervention, and 3 Months Post-Intervention
Likelihood to change their fat intake using the Stages of Change for Dietary Fat tool | Baseline, Immediately Post-Intervention, and 3 Months Post-Intervention
Likelihood to change their exercise using the Stages of Change for Physical Activity | Baseline, Immediately Post-Intervention, and 3 Months Post-Intervention
Change in diet quality using the Mediterranean Eating Pattern for Americans tool | Baseline and 3 Months Post-Intervention
Change in exercise status using the Exercise Vital Sign tool | Baseline and 3 Months Post-Intervention
Satisfaction with the educational intervention | Immediately Post-Intervention and 3 Months Post-Intervention
  Ordinal scale of 1 (very unsatisfied) to 7 (very satisfied)
New medications or changes in their anti-hypertensive medication use | 3 Months Post-Intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gottlieb, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No